CLINICAL TRIAL: NCT05348434
Title: Evaluation of Using 3D Printed Polyether Ether Ether Ketone Facial Implants in Repairing Maxillofacial Deformities
Brief Title: Evaluation of Using 3D Printed PEEK Facial Implants in Repairing Maxillofacial Deformities
Status: Completed | Type: Observational
Sponsor: Tishreen University (Other)
Responsible Party: Sponsor
Other Study IDs: Tishreen U- Maxillofacial sur
Record Dates: First submitted 2022-04-12; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Maxillofacial Trauma; Face Cancer; Mucormycosis
Keywords: facial implant; 3d printing; polyetheretherketone
MeSH Terms: conditions — Mucormycosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with maxillofacial deformities: 10 patients with maxillofacial deformities (trauma patients, war injuries, patients with pre-existing maxillofacial tumours, and meucrmycotic patients)
  Interventions: Procedure: 3D printed polyether ether ketone facial implants in repairing maxillofacial deformities

INTERVENTIONS:
Procedure: 3D printed polyether ether ketone facial implants in repairing maxillofacial deformities — All patients underwent Computed Tomography (CT) scans under the condition of providing a large number of slices (more than 200 slices) per axis, and the thickness of each slice is less than 1 mm with 64-bit resolution, Then the design of the required facial implant was carried out in coordination between the designer and the surgical team. The final form of the facial implant was printed from PolyEther Ether Ketone (PEEK), and then surgical work was performed for patients under general anaesthetic according to the appropriate surgical entrance. The implants were fixed in place using titanium screws
  Other Names: PSI PEEK

SUMMARY:
Objective: Evaluation of using 3D printed polyether ether ketone facial implants in repairing maxillofacial deformities.

Research materials and methods: The research sample consisted of 10 patients with facial deformities (maxillofacial trauma patients with hard tissue deficiencies, tumor patients who had previous facial surgery, patients have retrognathia, congenital malformation, patients with hemifacial microsomia - bone loss as a result of a mucormycotic infection or black fungus ) Between 2020 and 2021 in the Department of Oral and Maxillofacial Surgery in the Tishreen University Hospital - Latakia - Syria. All patients underwent Computed Tomography (CT) scans under the condition of providing a large number of slices (more than 200 slices) per axis, and the thickness of each slice is less than 1 mm with 64-bit resolution, Then the design of the required facial implant was carried out in coordination between the designer and the surgical team. The final form of the facial implant was printed from PolyEther Ether Ketone (PEEK), and then surgical work was performed for patients under general anaesthetic according to the appropriate surgical entrance. The implants were fixed in place using titanium screws and the patients were given appropriate pharmacological coverage .

DETAILED DESCRIPTION:
10 patients with maxillofacial deformities (trauma patients, war injuries, patients with pre-existing maxillofacial tumours, and mucormycotic patients) for reconstruction with 3D printed facial implants made of PEEK, between 2020 and 2021 in the Department of Oral and maxillofacial Surgery at the Tishreen University Hospital, Latakia, Syria. All patients underwent three-axial CT scan using a Toshiba Slice CT Scanner-Imaging, under the condition of providing a large number of slices (more than 200 slices) per axis, and the thickness of each slice is less than 1 mm with 64-bit resolution. Representative models of patient anatomical data were created based on the radiated raw data of the patient obtained via Digital Imaging and Communications in Medicine (DICOM) from the CT scan. The DICOM format is 0.3 to 0.6 mm thick, depending on the anatomical region. The medical modelling software (EXoCad) was used to compile DICOM data at the axial, sagittal, and coronal planes and then create a 3D virtual model of the anatomical region.

The surgeon and the manufacturing technician met to discuss the design format and any modifications required, with the proposed areas for placement of the titanium screws for the installation of the facial implant. The final default model for the facial implant was exported as a STereoLithography (STL) file and sent to the 3D printer, which was eventually made for the patient. The printer used in our study is a prototype of OO-Kuma Katana HT PEEK 3D Printer. After the process of printing, the facial implant is steam sterilized and then the implant is encapsulated. The surgical work of the patients was performed under general anaesthesia at the Tishreen University Hospital, Latakia, Syria, at the appropriate surgical entrance depending on the size and location of the deformity. The facial implant was checked to be suitable before stabilization and the required modifications were made during the process. The PSI was fixed in place using 1.5 to 2.0mm sized titanium screws, all patients received an intravenous 1.2g Augmentin dose and 0.5g of Flagyl during the procedure. After the surgery, patients received two doses of Augmentin, after which a prescription of Augmentin 1g and Flagyl 0.5g orally per day for a week was given.

ELIGIBILITY:
Inclusion Criteria:

- patients with facial deformities:

1. maxillofacial trauma patients with hard tissue deficiencies
2. tumor patients who had previous facial surgery
3. patients have retrognathia
4. congenital malformation
5. patients with hemifacial microsomia
6. bone loss as a result of a mucormycotic infection or black fungus

Exclusion Criteria:

1. acute stage oncology patients
2. There is not enough soft tissue to cover the facial implants

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients diagnosed with facial deformities at the Oral and Maxillofacial department of Tishreen University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of Cosmetic patients' satisfaction level . | after 3 months of the surgical procedure
  Three months after the surgery, we asked the patient to evaluate the aesthetic result by choosing a number from 1 to 5 , as 5 is the best cosmetic result.
  satisfaction scale :
  1. bad
  2. medium
  3. neutral
  4. satisfied
  5. very satisfied
Evaluation of infection after using 3D printed polyetheretherketone facial implants in repair of maxillofacial deformities | after surgical procedure a week, one month and three months
  A doctor _not included in the research team_ performed clinical examinations of patients after surgical procedure a week, one month and three months to check for clinical signs of infection .
  * When there are signs of infection, he records the number 1 .
  * When there are no signs of infection, he records the number 0 .

CONTACTS AND LOCATIONS:
Overall Officials: Hekmat Yacoub, PHD, Study Chair — Tishreen University; Ali Khalil, PHD, Study Director — Tishreen University; Ahmad Ahmad, Master, Principal Investigator — Tishreen University
Locations (1):
- Tishreen university, Latakia, Syria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Dua R, Rashad Z, Spears J, Dunn G, Maxwell M. Applications of 3D-Printed PEEK via Fused Filament Fabrication: A Systematic Review. Polymers (Basel). 2021 Nov 22;13(22):4046. doi: 10.3390/polym13224046. PMID 34833346
- [Result] Kang J, Zhang J, Zheng J, Wang L, Li D, Liu S. 3D-printed PEEK implant for mandibular defects repair - a new method. J Mech Behav Biomed Mater. 2021 Apr;116:104335. doi: 10.1016/j.jmbbm.2021.104335. Epub 2021 Jan 21. PMID 33494021
- [Result] Panayotov IV, Orti V, Cuisinier F, Yachouh J. Polyetheretherketone (PEEK) for medical applications. J Mater Sci Mater Med. 2016 Jul;27(7):118. doi: 10.1007/s10856-016-5731-4. Epub 2016 Jun 3. PMID 27259708